CLINICAL TRIAL: NCT07037264
Title: A Study of the Efficacy and Safety of Non-ablative Fractional Laser in the Treatment of Thyroidectomy Scars
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Medical Association (Network)
Responsible Party: Principal Investigator, Chengxin Li, Professor., Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2024-594-01
Record Dates: First submitted 2025-02-07; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Scars After Surgical Intervention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Non-ablative fractional laser treatment (Experimental)
  Interventions: Device: Non-ablative fractional laser treatment

INTERVENTIONS:
Device: Non-ablative fractional laser treatment — The entire scar area is sealed with local anesthetic for 60 minutes before laser treatment. Give the study side 1565 nm non-ablative fractional laser treatment, spot diameter 10～16 mm, energy 40～45 mJ/cm2, spot density 150～200/cm2,1~2passes.

SUMMARY:
The subject's neck thyroidectomy incision was bisected along the anterior midline. One side received 1565 nm non-ablative fractional laser treatment, designated as the study side, according to a computer-generated randomization scheme, while the other side received a sham treatment (the laser device emitted sound only, without delivering any energy), serving as the control side. Outcome indicators were recorded during follow-up, along with any related adverse events and/or reactions occurring during and after the treatment. The aim was to evaluate the effectiveness and safety of the 1565 nm non-ablative fractional laser in the treatment of postoperative thyroid scars.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is conscious, with no intellectual disability or cognitive difficulties, and understands and signs the informed consent form.
2. Healthy male and female subjects aged 18 to 70 years.
3. Fitzpatrick skin types I to V.
4. Women of childbearing age have used contraceptive measures within three months before enrollment.
5. The patient has undergone traditional thyroidectomy through the anterior neck approach within 15 days, with a surgical incision visible in the midline of the neck, symmetric along the anterior midline of the body surface; or the patient has undergone traditional thyroidectomy through the anterior neck approach within one year, with a linear hypertrophic surgical scar visible in the midline of the neck, symmetric along the anterior midline of the body surface.
6. The patient is able to comply with all the plans and requirements for visits, treatments, and assessments.requirements.

Exclusion Criteria:

1. Need for modified radical neck dissection or reoperation, or other surgical plans that may affect treatment and follow-up during the trial period;
2. Previous neck surgery;
3. Pregnant, planning to become pregnant during the study period, less than three months postpartum, or less than six weeks after completing breastfeeding;
4. History of keloid or delayed wound healing;
5. Uncontrolled systemic diseases;
6. History of mental disorders;
7. Presence of skin tumors or skin inflammation in the treatment area;
8. Active infection in the neck area or systemic infection;
9. Use of oral photosensitizing drugs or retinoids within six months before screening;
10. Use of anticoagulants, corticosteroids, immunosuppressants, or other drug treatments within three months before screening;
11. Exposure to strong ultraviolet radiation causing desquamation, erythema, or other conditions in the neck within one month before screening;
12. Participation in other drug/medical device clinical trials within one month before screening or planned participation during the study period;
13. Use of any other treatment methods for post-thyroidectomy scars except for silicone gel sheets and topical drugs before and during treatment;
14. Use of silicone gel sheets and topical drugs for post-thyroidectomy scars within seven days before starting treatment;
15. Patients allergic to compound lidocaine cream or its components, and no alternative to this drug is available;
16. Patients who, in the investigator's opinion, have other conditions that may affect compliance or are not suitable for participating in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The depth of scar echoes | Baseline,1month,2month,3month,4month,5month,8month,11month,17month
  Using the high-frequency skin ultrasound MD-300SⅡ, multiple-point measurements were taken in five different areas on both sides of the scar to determine the maximum and minimum values of scar echo depth and to calculate the average value of the five measurement points.The unit of measurement is millimeters.
The width of scar echoes | Baseline,1month,2month,3month,4month,5month,8month,11month,17month
  Using the high-frequency skin ultrasound MD-300SⅡ, multiple-point measurements were taken in five different areas on both sides of the scar to determine the maximum and minimum values of scar echo width and to calculate the average value of the five measurement points.The unit of measurement is millimeters.
Intensity of scar echoes | Baseline,1month,2month,3month,4month,5month,8month,11month,17month
  Using image processing software (Adobe Photoshop) to process the ultrasound images, the magic wand tool was used to select three areas of the same size on the scar. The average grayscale value of each area was read using the histogram function, and the average value of the five measurement points was calculated. The grayscale value is proportional to the echo intensity.
Modified vancouver scar scale score | Baseline,1month,2month,3month,4month,5month,8month,11month,17month
  The Modified Vancouver Scar Scale has a maximum score of 18 and a minimum score of 0, with higher scores indicating worse outcomes.

SECONDARY OUTCOMES:
Scar color | Baseline,1month,2month,3month,4month,5month,8month,11month,17month
  Using the multispectral microscopic imaging device (Multi view®) to perform multiple-point measurements in three different areas on both sides of the scar, calculate the grayscale and red concentration within a specific region, and separately calculate the average values of the three measurement points. The greater the average grayscale, the lighter the skin color, and vice versa. The higher the red concentration, the more severe the skin inflammation, and vice versa.
Scar area | Baseline,1month,2month,3month,4month,5month,8month,11month,17month
  Using the multispectral microscopic imaging device (Multi view®), identify the set of pixels with abrupt changes in brightness within the image, and employ edge detection algorithms to calculate the area of scars on both sides.
Patient and Observer Scar Assessment Scale score | Baseline,1month,2month,3month,4month,5month,8month,11month,17month
  The Patient and Observer Scar Assessment Scale consists of the Patient Scar Assessment Scale and the Observer Scar Assessment Scale. Both have a maximum score of 60 and a minimum score of 6, with higher scores indicating worse outcomes.
Manchester Scar Scale score | Baseline,1month,2month,3month,4month,5month,8month,11month,17month
  The Manchester Scar Scale has a maximum score of 28 and a minimum score of 5, with higher scores indicating worse outcomes.
Medical Outcomes Study Health Survey Short Form-36 Item score | Baseline,1month,2month,3month,4month,5month,8month,11month,17month
  Medical Outcomes Study Health Survey Short Form-36 Item (SF-36) consists of nine dimensions and 36 items, measuring eight aspects of health: Physical Functioning (PF), Role Limitations due to Physical Health (RP), Bodily Pain (BP), General Health Perceptions (GH), Vitality (VT), Social Functioning (SF), Role Limitations due to Emotional Problems (RE), and Mental Health (MH). Additionally, there is a self-assessment of health transition (HT) compared to health status one year ago, which is not included in the subscale or total scale scoring and reflects longitudinal dynamic changes. The scoring method involves calculating the sum of weighted item scores within each of the eight subscales to obtain the raw subscale scores, which are then transformed into standard scores ranging from 0 to 100. Higher scale scores indicate better quality of life.
Standardized assessment by doctor and patient | Baseline,1month,2month,3month,4month,5month,8month,11month,17month
  Two dermatologists on-site, two dermatologists via photographs, and the patient themselves answered standardized assessment questions, which included: Is there a difference between the left and right side scars? If "yes," which side is superior? The four dermatologists determined the final result using the following algorithm: If any of the four assessments indicated "no difference," or if the assessments of which half of the scar was superior did not match, the final result was determined to be "no difference."
Incidence of adverse events | Baseline,1month,2month,3month,4month,5month,8month,11month,17month
  Record and tally the frequency and severity of adverse events occurring during and after scar treatment.Incidence of adverse events = Number of cases with adverse events / Number of cases in the safety dataset × 100%.
Histological evaluation | 17month
  A 3 mm punch skin biopsy was taken from the center of the scar on both the study side and the control side. The biopsies underwent dewaxing, clearing, hematoxylin and eosin (HE) staining, Masson's trichrome staining, elastic fiber staining, and immunohistochemistry for matrix metalloproteinase (MMP9). The ImageJ software was used to calculate the average scar thickness in the HE-stained sections, the average area percentage of collagen fibers in the Masson's trichrome-stained sections, the average area percentage of elastic fibers in the elastic fiber-stained sections, and the average percentage of MMP9-positive cells on both sides.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA Genaral Hosptial, Beijing, Beijing Municipality, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT07037264/Prot_SAP_000.pdf
  • Informed Consent Form (2024-12-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT07037264/ICF_001.pdf